CLINICAL TRIAL: NCT04638192
Title: Design of Synchronized Pairing Peripheral Nerve Stimulation and Cortical Polarization to Promote Post-stroke Neuroplasticity for Hand Function Recovery
Brief Title: Transcranial Alternating Current Stimulation for Hand Function Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Chairman and Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017.663
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- subject-specific tACS (Experimental): Constant current (1mA) will be applied for 20min at subject-specific stimulation frequency and latency
  Interventions: Device: tACS
- standard tACS (Experimental): Constant current (1mA) will be applied for 20min at 20Hz with a fixed 25ms latency
  Interventions: Device: tACS
- Sham tACS (Sham Comparator): The stimulator will be shut down after 30s of stimulation. The patients will feel the initial itching sensation at the beginning in order to evaluate the placebo effect
  Interventions: Device: tACS

INTERVENTIONS:
Device: tACS — A pair of 25 cm2 rubber electrodes enclosed in saline-soaked sponges and affixed to the head with rubber bands.

SUMMARY:
tACS has the potential to directly induce cortical alterations in the intrinsic neural oscillation at specific frequencies, and the brain could mirror the induced frequencies of the external source of oscillations from the stimulation. Hence, tACS with matching stimulation frequency could be an effective means of enhancing brain oscillatory activity to potentially induce synaptic plasticity for restoration of damaged brain functions. However from the existing studies of applying tACS over the M1 in healthy and diseased brains, there is a wide range of applied stimulation frequencies and varied neuromodulation effects on motor behavior or cortical excitability at different frequencies. In this proposal, subject-specific stimulation frequency and latency will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis subsequent to first-ever unilateral stroke for more than 6 months;
* MCP and PIP finger joints can be extended to 180° passively;
* Sufficient cognition to follow the experimental instructions

Exclusion Criteria:

* Severe hand spasticity or hand deformity;
* History of alcohol or drug abuse or epilepsy;
* Bilateral brain infarcts;
* Severe cognitive deficits;
* Comprehensive aphasia;
* Contraindications to tACS and MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance imaging | 3-month after the 10th session training
  Structural and functional MRI

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 3-month after the 10th session training
  The ARAT has total 19 items, divided into 4 categories (grasp, grip, pinch, and gross arm movement). It ranges from 3 to 0 (best to worse).
Fugl-Meyer Assessment (Upper Extremity) | 3-month after the 10th session training
  The maximum score is 66, divided into 33 items in the form of a 3-point scale (0-2), 0 is cannot perform and 2 performs fully.
Wolf Motor Function Test (WMFT) | 3-month after the 10th session training
  The WMFT measures upper limb ability through timed and functional tasks. It has 17 items, ranging from 0 to 5 (worse to best).

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong